CLINICAL TRIAL: NCT02569229
Title: Glucose Tolerance and Its Clinical Impact in Children and Adolescents With Cystic Fibrosis
Brief Title: Glucose Tolerance in Children With Cystic Fibrosis
Acronym: GluTolCF
Status: Completed | Type: Observational
Sponsor: Christoph Saner (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor-Investigator, Christoph Saner, MD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: EKNZ 2015-143; KEK BE: 102/15 (Other: Ethics commitee of attending study site)
Record Dates: First submitted 2015-08-12; First posted 2015-10-06 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Glucose Intolerance; Cystic Fibrosis
Keywords: children; cystic fibrosis; glucose intolerance; continuous glucose measurement
MeSH Terms: conditions — Glucose Intolerance; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Glucose, C-Peptide, Insulin, HbA1c in blood specimen.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Cystic Fibrosis: Patients between 10-20 years of age with genetically determined cystic fibrosis followed at the university children's hospital Basel and university children's hospital Kinderklinik Bern, Switzerland. All patients will get the diagnostics for glucose tolerance with 3 different methods (CGMS, OGTT and optionally IVGTT).
  Interventions: Other: Diagnostics for glucose tolerance with 3 different methods.

INTERVENTIONS:
Other: Diagnostics for glucose tolerance with 3 different methods. — 1. A 7-day course of subcutaneous continuous glucose monitoring system (CGMS).
  2. An oral glucose tolerance test done within the 7 day period of CGMS.
  3. Optionally a intravenous glucose tolerance test done within the 7 day period of CGMS.

SUMMARY:
The aim is to describe the association of glucose tolerance measured with three different tools (continuous glucose measurement system - CGMS, oral glucose tolerance testing - OGTT and optional intravenous glucose tolerance testing -IVGTT) with parameters out of lung function and anthropometric parameters in patients with cystic fibrosis.

DETAILED DESCRIPTION:
Patients with cystic fibrosis (CF) with progressing disease are developing a glucose tolerance which resembles the metabolic state of a diabetic patient because of increasing impairment of endocrine pancreatic function. The prevalence of this diabetic metabolic state is increasing with age, reaching around 20% at the age of 20 years.

Over the last decade, research has already highlighted the negative influence of cystic fibrosis related diabetes (CFRD) on morbidity and mortality after the diagnosis of this condition.

As the deterioration in nutritional status and lung function can already be noticed 2-6 years before the onset of CFRD, the importance of early diagnosis in glucose abnormalities and its treatment therefore is crucial.

The currently used method to evaluate altered glucose metabolism in patients with CF is an annual oral glucose tolerance test (OGTT) with the glucose value after 120 min after oral ingestion of glucose-fluid as reference. This method may detect CFRD much later than we see deterioration of lung function and weight loss. This deterioration and the mortality in CF is related to CFRD.

An alternative diagnostic tool that has gained increasing attention and that is already routinely used in pediatric patients with diabetes mellitus type I is the continuous glucose monitoring system (CGMS) which was shown to be much more sensitive in detecting glucose abnormalities. To assess pancreatic endocrine dysfunction - the pathophysiologic cause for glucose intolerance - intravenous glucose tolerance testing (IVGTT) is the gold standard.

The investigator's aim is to describe the association of glucose tolerance measured with three different tools/assessment procedures (CGMS, OGTT and optional IVGTT) with lung function and anthropometric parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed cystic fibrosis aged between 10-20 years, under medical treatment at the University Children's Hospital Basel UKBB and at the University Children's Hospital, Inselspital Bern

Exclusion Criteria:

* Patients being under medical treatment with systemically administered glucocorticoid drugs or intravenously administered antibiotic treatment within 6 weeks before glucose tolerance testing.
* Patients with acute pulmonary exacerbation, defined by a pediatric pneumologist

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with genetically determined cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
% time spent above 8mmol/l, the area under the curve and the mean glucose value (in mmol/l) | Beginning at day 1, lasting 7 days
  These measurements will be gained out of the 7 day CGMS-course (continuous glucose monitoring system).
The glucose values given in mmol/l after 30', 60', 90' and 120 minutes during OGTT. | Within the 7 day course of CGMS
  Standard oral glucose tolerance test.
First phase insulin secretion and second phase insulin secretion out of IVGTT (intravenous glucose tolerance test). | Within the 7 day course of CGMS
  Standard intravenous glucose tolerance test.
FEV1% (forced expiratory volume at one second) out of the lung function testing | Within 3 months of the 7 day course of CGMS
Lung clearance index | Within 3 months of the 7 day course of CGMS
BMI-SDS (standard deviation score). | At day 1 of the CGMS course
HbA1c | Within the 7 day course of CGMS

SECONDARY OUTCOMES:
Comparing the performance between CGMS and OGTT related to clinical parameters. | 7 days
  The investigators compare the fit of a linear regression between the % time above 8mmol/l (out of CGMS) and the lung clearance index (LCI) with the fit of a linear regression of the 120min glucose value (out of OGTT) and the LCI. The same analysis will be performed comparing the fit of a regression between the % time above 8mmol/l (out of CGMS) and the FEV1% (out of lung function) with the fit of a linear regression of the 120min glucose value (out of OGTT) and the FEV1%. Finally, the same analysis will be performed comparing the fit of a linear regression using the % time above 8mmol/l (out of CGMS) and the BMI-SDS with the fit of a linear regression of the 120min glucose value (out of OGTT) and the BMI-SDS.

OTHER OUTCOMES:
Characterising glucose profiles over 24 hours | 7 days
  The investigators will describe computer-based modelling of the glucose curves obtained with the CGMS, aiming to describe inter-/ and intraindividual variability in the profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Saner, MD, Principal Investigator — University childrens Hospital, UKBB, Basel Switzerland; Urs Zumsteg, Prof, Study Director — University childrens Hospital, UKBB, Basel Switzerland
Locations (1):
- University childrens hospital Basel, UKBB, Basel, Switzerland